CLINICAL TRIAL: NCT03945071
Title: The Effect of Punctal Plugs in Reducing Ocular Surface Irritation After Povidone-Iodine Preparation of Intravitreal Injection
Brief Title: The Effect of Punctal Plugs on Ocular Surface After Povidone-Iodine Preparation of Intravitreal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 9810
Record Dates: First submitted 2019-02-10; First posted 2019-05-10 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Syndromes; Dry Eye; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Punctal Plugs

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Puntal plug (Active Comparator): Subjects will receive temporary punctal plug after intravitreal injection
  Interventions: Device: Punctal plug
- Non-Punctual plug (No Intervention): Subjects will not receive temporary punctal plug after intravitreal injection

INTERVENTIONS:
Device: Punctal plug — Punctal plug will be given to subjects after intravitreal injection in half of the study subjects
  Arms: Puntal plug

SUMMARY:
The aim of this study is to evaluate the effectiveness of punctal plugs in reducing ocular surface (eye surface) irritation after intravitreal injections prepared by povidone-iodine 5% solution.

DETAILED DESCRIPTION:
Intravitreal injection is a shot of medication into the eye. Many retinal diseases, such as diabetic retinopathy, neovascular age-related macular degeneration, and retinal vein occlusions require regular, periodic injections. Patients often reports eye surface irritation post intravitreal injection. One of the reasons for such discomfort is attributed to povidone-iodine solution used to clean the eye surface to reduce sight-threatening infections. Patients who already experience symptoms of dry eye are at increased risk of discomfort after povidone-iodine prepped intravitreal injections.

Povidone-iodine is known to be corrosive to the corneal epithelium and delay eye surface healing. Human tears contain proteins and chemicals that lubricate, heal, and protect the eye surface from infections and irritants. Adequate tear film therefore not only dilutes povidone-iodine, but also promotes corneal healing post povidone-iodine prepping.

The primary long-term objective of the present study is to investigate whether punctal plugs will reduce eye discomfort post intravitreal injections as reported by the Ocular Surface Disease Index (OSDI) and other relevant surveys. The secondary outcome is to describe any other risk and protective factors associated with eye surface discomfort after intravitreal injections.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of age-related macula degeneration
* Clinical diagnosis of diabetic retinopathy
* Clinical diagnosis of retinal vein occlusion

Exclusion Criteria:

* Currently wearing punctal plugs
* History of punctal cautery,
* Active ocular infection
* History of ocular infection
* Eyelid trauma
* Eyelid surgery
* Graft versus host disease
* Thyroid eye disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Change in ocular (eye) discomfort | From date of randomization until date of death from any cause, whichever came first, assessed up to 100 weeks
  Measure participants' level of discomfort after punctal plugs using the Ocular Surface Disease Index (OSDI), which is a paper survey that participants fill out based on their symptoms and level of ocular discomfort (if any).

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Shah, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Dean McGee Eye Institute, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Goldberg RA. How to prevent endophthalmitis after intravitreal injections. Int J Retina Vitreous. 2015 Aug 11;1:12. doi: 10.1186/s40942-015-0012-9. eCollection 2015. PMID 27847605
- [Background] Laude A, Lim JW, Srinagesh V, Tong L. The effect of intravitreal injections on dry eye, and proposed management strategies. Clin Ophthalmol. 2017 Aug 16;11:1491-1497. doi: 10.2147/OPTH.S136500. eCollection 2017. PMID 28860698
- [Background] Marcet MM, Shtein RM, Bradley EA, Deng SX, Meyer DR, Bilyk JR, Yen MT, Lee WB, Mawn LA. Safety and Efficacy of Lacrimal Drainage System Plugs for Dry Eye Syndrome: A Report by the American Academy of Ophthalmology. Ophthalmology. 2015 Aug;122(8):1681-7. doi: 10.1016/j.ophtha.2015.04.034. Epub 2015 May 30. PMID 26038339
- [Background] Ridder WH 3rd, Oquindo C, Dhamdhere K, Burke J. Effect of Povidone Iodine 5% on the Cornea, Vision, and Subjective Comfort. Optom Vis Sci. 2017 Jul;94(7):732-741. doi: 10.1097/OPX.0000000000001091. PMID 28609415
- [Background] Saedon H, Nosek J, Phillips J, Narendran N, Yang YC. Ocular surface effects of repeated application of povidone iodine in patients receiving frequent intravitreal injections. Cutan Ocul Toxicol. 2017 Dec;36(4):343-346. doi: 10.1080/15569527.2017.1291665. Epub 2017 Feb 28. PMID 28166657